CLINICAL TRIAL: NCT02921308
Title: Pulmonary Magnetic Resonance Imaging of Ex-preterm Children With and Without Bronchopulmonary Dysplasia To Understand Risk of Emphysematous Changes (PICTURE)
Brief Title: Pulmonary MRI of Ex-preterm Children With and Without BPD To Understand Risk of Emphysematous Changes
Acronym: PICTURE
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Sherri Katz, Pediatric Respirologist, Children's Hospital of Eastern Ontario
Other Study IDs: REB #16/31E
Record Dates: First submitted 2016-08-18; First posted 2016-10-03 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Prematurity; Bronchopulmonary dysplasia; MRI; PFT; Emphysema
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth; Emphysema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- With BPD: No intervention will be administered. After informed consent is obtained, children will undergo ultra-short echo time pulmonary MRI, followed by PFT and completion of questionnaires.
- Without BPD: No intervention will be administered. After informed consent is obtained, children will undergo ultra-short echo time pulmonary MRI, followed by PFT and completion of questionnaires.

SUMMARY:
Health Issue: Bronchopulmonary dysplasia (BPD), a chronic lung disease, is the most common complication of being born premature. Damage to the still developing lung stops the normal formation of the alveoli. Young adults with a history of BPD have lower lung function, early heart disease, and increased risk of death, compared to those without BPD. Recently, it has been reported that they may also develop a type of lung disease typically seen in older adults with a longstanding history of smoking. The severity of lung disease is usually measured using pulmonary function tests (PFT), but these tests may be normal, even in the presence of important changes in the fine structure of the lung. Such structural changes may be early markers of future lung disease and can be detected using lung magnetic resonance imaging (MRI). Unlike other ways of imaging the lungs, MRI does not expose people to harmful X-rays. To date, no studies have been done to examine the fine structure of the lung of school-aged children who had a history of BPD, to determine whether there are signs of lung disease that might not otherwise be obvious. This is important because once armed with this information, preventive measures can be taken to avoid worsening of lung disease.

Objective: 1) In 7-9 year-old children born extremely premature, lung MRI will be compared between those with and without BPD. The Investigators expect to observe more severe structural lung abnormalities in children with BPD, compared to those without BPD; 2) The Investigators will test to see if children with more severe MRI abnormalities also have worse lung function, and/or more symptoms of breathing problems. The Investigators expect to observe more PFT abnormalities in children with BPD than in those without and that these will match up with lung fine structure abnormalities identified on MRI.

How will work be undertaken? Children 7-9 years old who were born extremely prematurely will be recruited to participate in this study. Participants will be identified from Neonatal Follow-up clinics they attended. The Investigators will enroll 20 children with BPD and 20 without BPD. Participants will have lung MR images taken, during which they need to lie still for a few minutes. PFT will also be performed, during which they will blow into a machine. Parents will be asked to complete questionnaires about breathing problems, their living conditions (environment) and any doctor visits or hospital stays. Medical charts will be reviewed for information about their birth.

Unique/Innovative Aspects: This will be the first study using MRI as an innovative way to visualize and measure fine structure of the lung in children born prematurely with and without BPD. These findings may be early markers of lung disease, which would identify children who have, or are at risk of developing lung disease later in life, for whom the Investigators may be able to offer treatments now and/or prevent worsening of lung disease.

DETAILED DESCRIPTION:
Knowledge to Date: Bronchopulmonary dysplasia (BPD), the most common pulmonary complication of prematurity, occurs in 41% of infants born before 28 weeks' gestation.

Defined as a need for oxygen at 36 weeks' postmenstrual age,2 BPD results in longterm morbidity in children and adults, including reduced lung function, early cardiovascular disease and premature death The reported severity of such impairments varies, as studies have been conducted on small numbers of children with differing degrees of prematurity. Furthermore, it is unclear what markers are most sensitive to predict long-term respiratory compromise. While functional measures have been studied, micro-structural differences, that may be quantified using pulmonary magnetic resonance imaging (MRI), have not been evaluated in this population, and may provide earlier quantitative markers of future respiratory disease, including chronic obstructive pulmonary disease (COPD). Recent advances in the clinical care of preterm infants have permitted survival of ever more premature infants, in whom alveolar development is incomplete, representing a new, relatively unstudied and growing cohort with a new form of BPD.

This BPD is associated with arrested alveolar growth and development, with reduction in alveolar surface area and pulmonary capillary blood volume. Yet, little is known about the trajectory of associated lung changes through childhood. Traditional measures of pulmonary function are lower in school aged children with history of BPD than in those preterm-born without BPD, but they may still be within normal reference ranges. There is, however, evidence that pulmonary function declines more steeply between age 8-18 years in those with BPD and that lower infant lung function predicts lower adult lung function.

This is particularly concerning since there is increasing recognition that preterm born adults have a significant burden of early lung disease. Emphysema has been reported in young adults with a history of prematurity less extreme than the prematurity seen today. X-ray computed tomography (CT) imaging detects pulmonary abnormalities in 98%, with emphysema in 47% of this less premature cohort as young adults. Not all of those with CT abnormalities, however, have impaired pulmonary function tests (PFTs), thus highlighting the limitations of conventional PFTs to detect disease. In childhood, PFTs, while very powerful indicators of global lung health, may be relatively insensitive to detect early pulmonary structural changes and regional lung abnormalities. Pulmonary dysfunction may not cause symptoms at rest or correlate with PFTs in childhood, but may become apparent with exercise, infection, or aging. Structural changes in the lung parenchyma may already be present in childhood and may be earlier markers of current and future respiratory disease than conventional PFT. Such changes may be detected with pulmonary MRI of the lung, as has been shown in COPD and in pilot work in BPD MRI has significant advantages over CT, including lack of exposure to ionizing radiation and high resolution of fine tissue structure. Recent advances in pulmonary MRI, including ultra-short echo time pulse sequences, generate pulmonary images with enhanced parenchymal signal intensity which rival CT images for visualization of lung parenchyma and vasculature. MRI is emerging as a research tool and may ultimately replace CT for pediatric thoracic imaging tasks and serial evaluations.

To the Investigators knowledge, conventional and ultra-short echo time 1H MRI studies of children with histories of prematurity and BPD have not been performed to quantify microstructural pulmonary abnormalities. The Investigators therefore propose a study to compare pulmonary micro-structural (MRI) and functional (PFT) abnormalities in premature children with and without history of BPD. The investigators hypothesize that pulmonary tissue destruction and/or emphysematous changes will be evident on MRI and will be worse in ex-premature infants with a history of BPD than in those without history of BPD. Further, the investigators hypothesize that MRI will be more sensitive to detect lung changes than PFT, but that MRI changes will correlate with PFT abnormalities. Ultimately, this information will form the basis of future longitudinal studies to evaluate progression of pulmonary disease and assess effects of new treatment strategies in this population.

Research Questions Amongst 7-9 year old children with a history of prematurity (< 28 weeks' gestation), comparing those with and without a history of BPD

1. Are there measureable differences in pulmonary micro-structure, quantified using MRI signal intensity (primary question)?
2. What is the association between pulmonary micro-structural measurements quantified using pulmonary MRI and pulmonary function outcomes (secondary questions):

   1. airflow limitation, as measured by forced expiratory volume in one second (FEV1), FEV1/FVC, mid-expiratory flows (FEF25-75)
   2. lung volumes and gas trapping , as measured by total lung capacity (TLC), residual volume (RV) and RV/TLC ratio
   3. diffusion capacity of carbon monoxide (DLCO), a marker of pulmonary alveolar volume and pulmonary diffusing capacity
   4. respiratory symptoms, social and environmental exposure history and healthcare utilization, assessed by validated questionnaire (ATS-DLD-78-a) Methods Study Setting: This cross-sectional study will be carried out at three Canadian tertiary care pediatric centres (Children's Hospital of Eastern Ontario, Ottawa, Ontario, The Hospital for Sick Children, Toronto, Ontario and Centre Hospitalier Universitaire (CHU) Sainte-Justine, Montreal, Quebec). Ethics approval will be obtained at all participating sites. Analysis: Descriptive statistics will be used to describe the two groups. The primary analysis will be a comparison of signal intensity between children with a history of BPD and those without, adjusting for exposure to earlier (24-26 weeks) or later (27-28 weeks) gestational age, using a two-way analysis of variance. Secondary analyses will examine the association between MRI signal intensity and PFT, as well as signal intensity and respiratory symptoms from the ATS-DLD-78-c questionnaire, using Spearman correlations. Exploratory analyses will also examine the association between PFT and respiratory symptoms, as well as parental smoking exposure, the relationship of obstetrical and neonatal historical factors to signal intensity, PFT, and respiratory symptoms.

Feasibility: Imaging Feasibility: The MRI pulse sequence that is the foundation for this study was previously developed and validated at 3T on a GE scanner by Dr. Parraga, who serves as Co-Principal Investigator of this proposed research.42 The MR acquisitions will be enabled using MR infrastructure at all 3 sites and 32 channel cardiac coils. Proof-of-concept for the presence of extensive emphysema is provided for a 25 year old with a history of prematurity and BPD, with significant MRI-evidence of widespread alveolar and acinar duct abnormalities that are consistent with emphysema Recruitment Feasibility: Each year, approximately 400 infants born < 28 weeks' gestation attend neonatal clinic follow-up visits at 18 months of age, at the three participating centres. As there are already established databases of these children at each site, identification of those eligible for study participation will be easily achieved.

At CHU Sainte-Justine, approximately 80 children aged 5-7 years are seen annually and from a previous study recruiting at 5 years, participation rate was 60%, further supporting feasibility for this study. Anticipated Results and Conclusions The Investigators anticipate that there will be significantly more severe pulmonary micro-structural abnormalities, as evidenced by lower pulmonary mean signal intensity, in 7-9 year olds born at less than 28 weeks' gestation, with a history of BPD, as compared to children born at less than 28 weeks' gestation without BPD. The investigators expect that mean MRI-derived signal intensity will correlate significantly with PFT measurements, as well as with the presence of chronic respiratory symptoms and increased healthcare utilization. This is the first study using innovative MRI techniques in relation to functional testing that will help characterize regional pulmonary tissue destruction and/or emphysematous changes present in children with a history of extreme prematurity, with and without BPD. In particular, MRI measurements may be more sensitive markers of early lung disease than PFT or respiratory symptoms. Since these children may only manifest signs of respiratory impairment in the presence of stressors, knowledge of these MRI changes may prompt earlier or more aggressive respiratory support and treatment to prevent respiratory compromise. Ultimately, there may be opportunity in future to intervene with additional treatments that may halt progression to adult lung disease. This is particularly important, given the increasing body of evidence for early COPD-like disease in this group. This work may identify a BPD-COPD overlap syndrome, with unique pathophysiology and potentially differential response to treatments from traditional COPD.

Potential Challenges: Children will be recruited for this study from neonatal follow-up clinic databases that capture all of those graduating from the neonatal nursery and surviving to 18 months. It is possible that some families may have since relocated or have been lost to follow-up and/or that those willing to participate in a research study at age 7-9 years will differ from those not willing/able to participate. Further, by studying children able to perform PFT and to cooperate for MRI, the investigators will exclude those with significant neurodevelopmental delay, who may also have more severe lung disease. As these are the main study outcomes, however, this will be necessary. Inclusion of children with a history of BPD ensures that those at the more severe end of the spectrum of early pulmonary complications, who are expected to have more severe lung disease, are studied. Exercise testing is another methodology to assess pulmonary and cardiovascular function. It is beyond the feasibility and budget ($200 per test) for this study and also requires coordination tasks that may be challenging for some participants. Nonetheless, it is an important consideration for future work. There are few precedents for pulmonary MRI in children, particularly in those with prematurity and BPD. Traditionally, MRI has been considered suboptimal in comparison to CT for lung parenchyma imaging, due to the low tissue density and loss of signal from magnetic field inhomogeneity at the air lung interfaces. Novel ultra-short echo time (UTE) pulse sequences, however, permit greater signal from the pulmonary parenchyma, which makes MRI a viable strategy to assess emphysematous changes in this population, without exposure to ionizing radiation. In the neonatal intensive care unit, MRI has shown signal decreases suggestive of alveolar simplification (emphysema) in those with severe BPD. It is possible that children with a history of extreme prematurity without BPD will also have some degree of pulmonary parenchymal change on MRI, although it is still expected that abnormalities will be more severe in those with a history of BPD. This study is, however, powered to detect smaller differences in signal intensity between groups than observed in adult COPD studies. The investigators are not using a healthy term control group because the purpose of this research is to assess radiological and functional biomarkers that will help clinicians and researchers identify among preterm born children those at greater risk of long-lasting pulmonary problems who would benefit the most from treatment.

Relevance: The ever growing population of extremely preterm born individuals, representing approximately 27,000 Canadians less than 18 years old, of whom approximately 40% have BPD, is at risk of development of early COPD-like emphysematous changes. Thus, neonatal conditions may be at the origin of a substantial and disproportionately high burden of adult lung disease, associated with significant morbidity and mortality. Prematurity and BPD, in addition to smoking, is one of the strongest predictors of obstructive airways disease in later life. In order to promote lung health and reduce the global burden of chronic lung disease, it is necessary to understand the trajectory of lung growth, development and decline across the lifespan in this at-risk population. Use of novel imaging strategies, more sensitive than PFT or respiratory symptoms to quantify early changes in the lung, provides new knowledge about the natural history of BPD in this population. Furthermore, MRI changes can quantify improvement associated with therapeutic interventions and can be safely serially evaluated across the lifespan. This is particularly important and exciting, given new therapies on the horizon to treat BPD, including stem cell treatments.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria: Children born pre-term at less than 28 weeks' gestation, currently aged 7-9 years, with and without BPD will be included.

Exclusion Criteria:

* Children with known interstitial lung disease, congenital lung anomalies, cystic fibrosis, ciliary dysfunction, immunodeficiency, neuromuscular disease or structural heart disease, which may have associated PFT and/or MRI findings;
* Genetic syndromes which may have other associated structural lung anomalies;
* Any contraindications for MRI;
* Severe neurosensory deficits which would prevent test completion;
* Viral or bacterial respiratory infection within 6 weeks.50

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children born pre-term at less than 28 weeks' gestation, currently aged 7-9 years, with and without BPD will be included. BPD will be defined as need for oxygen at 36 weeks' postmenstrual age,2 which includes those with moderate-severe disease.47 Children 7-9 years of age were selected in order to include the youngest age at which pulmonary function, including lung volumes and single breath pulmonary diffusing capacity for carbon monoxide, can routinely be reliably measured using methods that require subject cooperation.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

PRIMARY OUTCOMES:
Primary Outcome: MRI-derived Pulmonary Microstructure measurements | Assessed at one time point at Baseline
  Images will be acquired in 10-15 seconds in all subjects using a 2D radial ultra-short echo time pulse sequence, to quantify signal intensity as a surrogate of parenchymal tissue density. Subjects will be asked to breath normally and then inhale a fixed volume of air from functional residual capacity (the volume of which is calibrated to 50% of inspiratory capacity) and hold their breath while images are acquired, as previously described. The pulse sequence for imaging will be developed as previously described and validated for the different MR scanner platforms at the three participating sites, through the Imaging platform of the Canadian Respiratory Research Network. All image volumes will be scaled to functional residual capacity plus 50% of inspiratory capacity and will be acquired in breath-hold at that inspiratory volume. The CRRN Imaging platform will also provide test objects for calibration of 1H MRI signal intensity to ensure

SECONDARY OUTCOMES:
Height | Assessed at one time point at Baseline
  Height and weight will be measured at baseline prior to doing the Pulmonary Function Testing. It is important to have current measurements of Height and weight as they are used in the calculation of some of the variables that are measured during PFTs
Weight | Assessed at one time point at Baseline
  Height and weight will be measured at baseline prior to doing the Pulmonary Function Testing. It is important to have current measurements of Height and weight as they are used in the calculation of some of the variables that are measured during PFTs
Airflow limitations | Assessed at one time point at Baseline
  Outcomes related to airflow limitation, including FEV1, was selected as it has been shown in previous studied to be reduced in children and adults with a history of prematurity and BPD,
Airflow limitations | Assessed at one time point at Baseline
  Outcomes related to airflow limitation, including FEV1/FVC was selected as it has been shown in previous studied to be reduced in children and adults with a history of prematurity and BPD,
Airflow limitations | Assessed at one time point at Baseline
  Outcomes related to airflow limitation, including mid-expiratory flows (FEF), was selected as it has been shown in previous studied to be reduced in children and adults with a history of prematurity and BPD,
Spirometry pre and post bronchodilators | Assessed at one time point at Baseline
  Spirometry pre and post bronchodilators, lung volumes will be performed on all participants, according to established American Thoracic Society criteria for test performance and scoring. Published predictive equations for spirometry, lung volumes and DLCO will be used. Lung volumes, assessed by TLC, RV and RV/TLC ratio, will be used to identify gas trapping and will be correlated with gas trapping and ventilation inhomogeneity on MRI.
Lung Volumes - Total Lung Capacity | Assessed at one time point at Baseline
  Spirometry pre and post bronchodilators, lung volumes will be performed on all participants, according to established American Thoracic Society criteria for test performance and scoring. Published predictive equations for spirometry, lung volumes and DLCO will be used. Lung volumes, assessed by TLC, RV and RV/TLC ratio, will be used to identify gas trapping and will be correlated with gas trapping and ventilation inhomogeneity on MRI.
Lung Volumes - Residual Volume | Assessed at one time point at Baseline
  Spirometry pre and post bronchodilators, lung volumes will be performed on all participants, according to established American Thoracic Society criteria for test performance and scoring. Published predictive equations for spirometry, lung volumes and DLCO will be used. Lung volumes, assessed by TLC, RV and RV/TLC ratio, will be used to identify gas trapping and will be correlated with gas trapping and ventilation inhomogeneity on MRI.
Lung Volumes - RV/TLC ratio | Assessed at one time point at Baseline
  Spirometry pre and post bronchodilators, DLco will be performed on all participants, according to established American Thoracic Society criteria for test performance and scoring. Published predictive equations for spirometry, lung volumes and DLCO will be used. Lung volumes, assessed by TLC, RV and RV/TLC ratio, will be used to identify gas trapping and will be correlated with gas trapping and ventilation inhomogeneity on MRI.
DLCO | Assessed at one time point at Baseline
  Spirometry pre and post bronchodilators, DLco will be performed on all participants, according to established American Thoracic Society criteria for test performance and scoring. Published predictive equations for spirometry, lung volumes and DLCO will be used. Lung volumes, assessed by TLC, RV and RV/TLC ratio, will be used to identify gas trapping and will be correlated with gas trapping and ventilation inhomogeneity on MRI.
Diffusion capacity | Assessed at one time point at Baseline
  Diffusion capacity was included as an outcome, as this may be a sensitive marker of alveolar simplification, a hallmark of the "new" BPD.
Medical History | Assessed once from the Canadian Neonatal Network database
  Additional information necessary to describe the population's obstetrical and neonatal history will be obtained from data already abstracted in the Canadian Neonatal Network database, which covers the time frame of birth to the present time, to which all centers have access, and through review of the medical charts, including: (1) Maternal data: prenatal corticosteroids, chorioamnionitis; (b) Neonatal data: gestational age, birth weight, APGAR, respiratory-related treatment (surfactant, mechanical ventilation, oxygen, steroids), medical complications (sepsis, patent ductus).
ATS-DLD-78-c | Assessed at one time point at Baseline
  A validated questionnaire (ATS-DLD-78-c) will be administered to collect information on respiratory symptoms and the following determinants of health: (1) Socio-economic status, occupation and education level of parents. (2) Family history of chronic pulmonary diseases; (3) Environmental exposures: cigarette smoke, pets, wood stove, daycare/school, living quarters; (4) Personal medical history: hospitalization for respiratory-related illness and current medication use.
MODIFIED EPWORT SLEEPINESS SCALE | Assessed at one time point at Baseline
  On the night of the sleep study the patients will be provided with a sleep questionnaire designed to elicit a history of sleep-disordered breathing, Excessive daytime sleepiness is considered present if the Epworth score is ≥ 11.14
Pediatric Sleep Questionnaire (Chervin); | Assessed at one time point at Baseline
  On the night of the sleep study the patients will be provided with a sleep questionnaire (developed by Chervin et al) designed to elicit a history of sleep-disordered breathing, SDB will be considered present if 8 of Chervin's questions are positive.
The Habitual Activity Estimation Scale (HAES) | Assessed at one time point at Baseline
  The HAES questionnaire will be administered at baseline to assess the level of physical activity of the child. This validated questionnaire has been used in many clinical populations of children(149;150) and captures both the duration and intensity of physical activity.(151;152) Information is completed on one typical weekday and one weekend day. The questionnaire takes approximately 15 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Sherri Katz, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (4):
- Canada (4):
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Children"s Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - CHU-Sainte Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Katz SL, Parraga G, Luu TM, Santyr G, Abdeen N, Deschenes S, Tse SM, Couch MJ, Barrowman N, Hayawi L, Momoli F, Blinder H, Thebaud B, Nuyt AM, Ben Fadel N, Moraes TJ. Pulmonary Magnetic Resonance Imaging of Ex-Preterm Children with and without Bronchopulmonary Dysplasia. Ann Am Thorac Soc. 2022 Jul;19(7):1149-1157. doi: 10.1513/AnnalsATS.202106-691OC. PMID 35030070